CLINICAL TRIAL: NCT06737172
Title: Cross-sectional Analysis of Functional and Structural Outcomes in Children, Adolescents and Young Adults Within Follow-up of Bone or Soft Tissue Sarcomas of the Lower Extremity
Brief Title: Functional and Structural Outcomes Following Childhood Bone or Soft Tissue Sarcomas of the Lower Extremity
Acronym: FOCUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other)
Responsible Party: Principal Investigator, Sabine Kesting, Head of Pediatric Exercise Oncology Working Group, Technical University of Munich
Other Study IDs: FOCUS
Record Dates: First submitted 2024-11-25; First posted 2024-12-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Soft Tissue Sarcoma of the Lower Extremity; Bone Sarcoma of the Lower Extremity; Childhood and Adolescent Cancer
Keywords: bone tumor; soft tissue sarcoma; functional outcomes; cross-sectional analysis
MeSH Terms: conditions — Bone Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survivors of childhood bone or soft tissue sarcomas of the lower extremity: Survivors aged 6-18 years who were treated for bone or soft tissue sarcoma of the lower extremity in one of the recruiting study sites, 1-5 years following the end of therapy

SUMMARY:
Soft tissue and bone sarcomas of the lower extremity pose significant challenges for affected individuals, often associated with considerable burden. Chemotherapy, load restrictions, and surgery frequently result in long-term physical limitations, causing structural and functional deterioration. These challenges are particularly pronounced in childhood and adolescence, as they affect physiological development, resilience, and autonomy. Yet, it remains unclear whether these deficits can be fully compensated after treatment or if they result in long-term limitations, as this has not been sufficiently studied.

This bicentric study includes children and adolescents undergoing follow-up care for soft tissue or bone sarcoma of the lower extremity within 1 to 5 years since end of therapy. The cohort did not receive any specific prehabilitative training during neoadjuvant therapy. Participants will be divided into two subgroups based on the study site: (1) participants who participated in a non-specific exercise program during acute therapy and (2) participants who did not receive any exercise promotion during acute therapy. Target sample size is n=16. The study has been consented by the local ethics committee.

Several structural and functional parameters are measured to document the natural status of muscular structures and functional abilities after the treatment of a solid tumor in the lower extremities, with a focus on identifying specific deficits and the associated long-term limitations in daily life. The measurements include psoas muscle area, body composition, strength, mobility, balance ability, gait analysis, two questionnaires on physical activity and quality of life, and quantitative measures of the clinical course during acute treatment (days of hospitalization, infection rates, etc.).

For children and adolescents, daily functionality and the experience of autonomy are crucial for physiological development and contribute significantly to quality of life. Therefore, these factors should be investigated and supported in this cohort, a group that is currently underrepresented in scientific research.

ELIGIBILITY:
Inclusion Criteria:

* Cessation of treatment for a bone tumor or soft tissue sarcoma of the lower extremity 1-5 years ago
* Age Range of 6 to 18 years
* Treatment has been conducted at one of the two designated study sites

Exclusion Criteria:

* Medical contraindications for testing (e.g. injury, pain, dizziness, lack of orthopedic clearance for weight-bearing in the tumor region, other acute orthopedic limitations unrelated to the underlying condition, etc.)
* Language barriers that prevent understanding of the instructions for study participation
* Cognitive impairment or developmental delay that hinders comprehension of the instructions in the testing situation, thereby preventing standardized diagnostic data collection

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants include children and adolescents during follow-up in Munich/Germany for soft tissue sarcoma or bone tumor at the lower extremity currently 1-5 years after cessation of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Total psoas muscle area | At diagnostic procedure 1-5 years following the end of therapy
  Total psoas muscle area at lumbal level (L4) analyzed via MRI or PET CT

SECONDARY OUTCOMES:
Fat-free mass | At diagnostic procedure 1-5 years following the end of therapy
  The weight of all body components excluding fat, measured in kilograms, using bioimpedance analysis.
  Outcome measures 2.-6. will be combined to report body composition.
Fat mass | At diagnostic procedure 1-5 years following the end of therapy
  Total body fat weight, measured in kilograms, assessed via bioimpedance analysis.
  Outcome measures 2.-6. will be combined to report body composition.
Total body water | At diagnostic procedure 1-5 years following the end of therapy
  The proportion of total body water in kg, expressed as percentage, measured through bioimpedance analysis.
  Outcome measures 2.-6. will be combined to report body composition.
Body cell mass | At diagnostic procedure 1-5 years following the end of therapy
  The mass of metabolically active cells in the body, measured in kilograms, via bioimpedance analysis.
  Outcome measures 2.-6. will be combined to report body composition.
Phase angle | At diagnostic procedure 1-5 years following the end of therapy
  An indicator of cellular health and membrane integrity, measured in degrees using bioimpedance analysis.
  Outcome measures 2.-6. will be combined to report body composition.
Muscle strength | At diagnostic procedure, 1-5 years following the end of therapy
  Overall muscle strength measured by hand-grip dynamometry.
Range of motion of the adjacent joints | At diagnostic procedure, 1-5 years following the end of therapy
  Range of motion of the adjacent joints measured with an analog goniometer.
Gait analysis | At diagnostic procedure, 1-5 years following the end of therapy
  Gait analysis measured with a force plate to analyze how pressure is distributed during stance phases of walking (vertical ground reaction force during loading response, mid stance, terminal stance, toe off).
Path length | At diagnostic procedure 1-5 years following the end of therapy
  The total distance traveled by the center of pressure during balance assessment, measured in centimeters using a force plate. Outcome measures 10.-13. will be combined to report balance ability.
Mean velocity | At diagnostic procedure 1-5 years following the end of therapy
  The average speed of center of pressure shifts during balance assessment, measured in meters per second with a force plate. Outcome measures 10.-13. will be combined to report balance ability.
Sway angle | At diagnostic procedure 1-5 years following the end of therapy
  The angular deviation of the center of pressure from a neutral position during balance tasks, measured in degrees using a force plate. Outcome measures 10.-13. will be combined to report balance ability.
Equlibrium score | At diagnostic procedure 1-5 years following the end of therapy
  Calculated from the anterior-posterior and medial-lateral projection of the 90% Standard Ellipse and estimated height of center of gravity during balance tasks in percentage using a force plate. Outcome measures 10.-13. will be combined to report balance ability.
Level of physical activity | At diagnostic procedure, 1-5 years following the end of therapy
  Level of physical activity following therapy measured with the standardized ActiOn questionnaire
Quality of life | At diagnostic procedure, 1-5 years following the end of therapy
  Quality of life during and following therapy measured with the standardized and validated KINDL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sabine V Kesting, Dr. rer. medic., Principal Investigator — Technical University of Munich; Irene von-Luettichau, Prof. Dr. med., Principal Investigator — Technical University of Munich
Locations (2):
- Germany (2):
  - Dr. von Haunersches Kinderspital, University of Munich, Munich, Bavaria
  - Technical University of Munich, Germany; TUM School of Medicine and Health, Department of Pediatrics. German Center for Child and Adolescent Health (DZKJ), partner site Munich, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basteck S, Guder WK, Dirksen U, Krombholz A, Streitburger A, Reinhardt D, Gotte M. Effects of an Exercise Intervention on Gait Function in Young Survivors of Osteosarcoma with Megaendoprosthesis of the Lower Extremity-Results from the Pilot Randomized Controlled Trial proGAIT. Curr Oncol. 2022 Oct 14;29(10):7754-7767. doi: 10.3390/curroncol29100613. PMID 36290890
- [Background] Bhagat A, Kleinerman ES. Anthracycline-Induced Cardiotoxicity: Causes, Mechanisms, and Prevention. Adv Exp Med Biol. 2020;1257:181-192. doi: 10.1007/978-3-030-43032-0_15. PMID 32483740
- [Background] Ehrhardt MJ, Leerink JM, Mulder RL, Mavinkurve-Groothuis A, Kok W, Nohria A, Nathan PC, Merkx R, de Baat E, Asogwa OA, Skinner R, Wallace H, Lieke Feijen EAM, de Ville de Goyet M, Prasad M, Bardi E, Pavasovic V, van der Pal H, Fresneau B, Demoor-Goldschmidt C, Hennewig U, Steinberger J, Plummer C, Chen MH, Teske AJ, Haddy N, van Dalen EC, Constine LS, Chow EJ, Levitt G, Hudson MM, Kremer LCM, Armenian SH. Systematic review and updated recommendations for cardiomyopathy surveillance for survivors of childhood, adolescent, and young adult cancer from the International Late Effects of Childhood Cancer Guideline Harmonization Group. Lancet Oncol. 2023 Mar;24(3):e108-e120. doi: 10.1016/S1470-2045(23)00012-8. Epub 2023 Feb 14. PMID 37052966
- [Background] Furtado S, Errington L, Godfrey A, Rochester L, Gerrand C. Objective clinical measurement of physical functioning after treatment for lower extremity sarcoma - A systematic review. Eur J Surg Oncol. 2017 Jun;43(6):968-993. doi: 10.1016/j.ejso.2016.10.002. Epub 2016 Oct 14. PMID 27836415
- [Background] Garcia MB, Ness KK, Schadler KL. Exercise and Physical Activity in Patients with Osteosarcoma and Survivors. Adv Exp Med Biol. 2020;1257:193-207. doi: 10.1007/978-3-030-43032-0_16. PMID 32483741
- [Background] Gauss G, Beller R, Boos J, Daggelmann J, Stalf H, Wiskemann J, Gotte M. Adverse Events During Supervised Exercise Interventions in Pediatric Oncology-A Nationwide Survey. Front Pediatr. 2021 Aug 19;9:682496. doi: 10.3389/fped.2021.682496. eCollection 2021. PMID 34490156
- [Background] Gotte M, Gauss G, Dirksen U, Driever PH, Basu O, Baumann FT, Wiskemann J, Boos J, Kesting SV. Multidisciplinary Network ActiveOncoKids guidelines for providing movement and exercise in pediatric oncology: Consensus-based recommendations. Pediatr Blood Cancer. 2022 Nov;69(11):e29953. doi: 10.1002/pbc.29953. Epub 2022 Sep 8. PMID 36073842
- [Background] Lurz E, Patel H, Lebovic G, Quammie C, Woolfson JP, Perez M, Ricciuto A, Wales PW, Kamath BM, Chavhan GB, Juni P, Ng VL. Paediatric reference values for total psoas muscle area. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):405-414. doi: 10.1002/jcsm.12514. Epub 2020 Jan 9. PMID 31920002
- [Background] Pilz F, Vill K, Rawer R, Bonfert M, Tacke M, Heussinger N, Muller-Felber W, Blaschek A. Mechanography in children: pediatric references in postural control. J Musculoskelet Neuronal Interact. 2022 Dec 1;22(4):431-454. PMID 36458382
- [Background] Runco DV, Zimmers TA, Bonetto A. The urgent need to improve childhood cancer cachexia. Trends Cancer. 2022 Dec;8(12):976-979. doi: 10.1016/j.trecan.2022.07.005. Epub 2022 Aug 3. PMID 35931609
- [Background] Winter CC, Muller C, Hardes J, Gosheger G, Boos J, Rosenbaum D. The effect of individualized exercise interventions during treatment in pediatric patients with a malignant bone tumor. Support Care Cancer. 2013 Jun;21(6):1629-36. doi: 10.1007/s00520-012-1707-1. Epub 2013 Jan 5. PMID 23292667